CLINICAL TRIAL: NCT05022576
Title: Trans Gluteal Automated Robotic Arm Assisted Ga-68 Prostate-specific Membrane Antigen Position Emission Tomography/ Computed Tomography Guided Percutaneous Prostate Biopsies.
Brief Title: Robotic-arm Assisted Ga-68 PSMA PET/CT Guided Transgluteal Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajender Kumar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INT/IEC/2019/001994
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
Keywords: Positron Emission Tomography Computed Tomography; Glu-NH-CO-NH-Lys-(Ahx)-((68)Ga(HBED-CC)); Biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA PET/CT guided biopsy arm (Experimental): Ga-68 PSMA PET/CT imaging is now routinely done in patients with prostate cancer with biochemical recurrence, response evaluation and even in patients with clinical suspicion of prostate cancer. In the present study, we aim to plan robotic arm-assisted Ga-68 PSMA guided transgluteal prostatic biopsies.
  Interventions: Diagnostic Test: Robotic arm assisted PSMA PET/CT guided prostate biopsy

INTERVENTIONS:
Diagnostic Test: Robotic arm assisted PSMA PET/CT guided prostate biopsy — The patients were positioned prone on PET/CT table. The regional PET/CT image of the lower pelvic region were acquired for the procedure. The images were transferred to the ROBIO™ EX workstation. The ARA workstation determined the needle trajectory, depth of the lesion and angulations. The planned trajectory was appraised for its relationship with the vital organs. Strict surgical aseptic approach was followed for the procedure under local anesthesia. An 18G x 20cm coaxial system was manually introduced through the bush and pushed with the help of robotic arm through the gluteal skin entry site to the predetermined depth in the prostate. The real-time placement of the needle was confirmed with low dose CT and the biopsy specimens were retrieved. After the procedure, patient vitals and any difficulty in micturition were observed for two hours in the recovery area. The specimens were sent for histopathological examination.

SUMMARY:
Gallium-68 prostate-specific-membrane-antigen (Ga-68 PSMA) PET/CT is being used in Prostate cancer imaging. In the present study, we aimed to evaluate the efficacy and safety of robotic arm-assisted Ga-68 PSMA PET/CT-guided transgluteal prostatic biopsy.

Seventy-eight participants with a clinical suspicion of PCa were recruited from January 2019 to September 2020. All the patients underwent whole-body Ga-68 PSMA PET/CT. The patients with PSMA-avid lesion in the prostate underwent robotic arm-assisted PET-guided transgluteal biopsies. The degree of pain during the procedure, procedure-related complications and histopathology were evaluated.

ELIGIBILITY:
Inclusion Criteria:

i. Clinically or biochemically suspected cases of Ca Prostate. ii. Patients with PSMA avid lesion in the prostate iii. Patients, who were ready to give written informed consent for biopsy iv. In good general condition (Karnofsky performance status, KPS, of more than 70).

Exclusion Criteria:

i. No focal PSMA expressing lesion in the prostate ii. Patients who refused to give written informed consent iii. Abnormal coagulation profile iv. Acute prostatitis, any severe acute or chronic medical condition

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Evaluation of patients with clinically suspected prostate cancer which is applicable to male patients only
Enrollment: 78 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
The diagnostic yield of the procedure | three months
  Obtaining a biopsy specimen from the PSMA expressing site of the prostate in patients with clinical suspicion of prostate cancer to establish a pathological diagnosis.
Safety of the procedure | Seven days
  The periprocedural and post procedural adverse effects were documented

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be obtained directly from the principal investigator on reasonable request.

REFERENCES:
- [Derived] Kumar R, Singh SK, Mittal BR, Vadi SK, Kakkar N, Singh H, Krishnaraju VS, Kumar S, Bhattacharya A. Safety and Diagnostic Yield of 68Ga Prostate-specific Membrane Antigen PET/CT-guided Robotic-assisted Transgluteal Prostatic Biopsy. Radiology. 2022 May;303(2):392-398. doi: 10.1148/radiol.204066. Epub 2022 Feb 22. PMID 35191735